CLINICAL TRIAL: NCT01317992
Title: Ibudilast in the Treatment of Medication Overuse Headache: A Double-blind, Randomised, Placebo-controlled Pilot Study
Brief Title: Ibudilast in the Treatment of Medication Overuse Headache
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Collaborators: University of South Australia (Other)
Responsible Party: Principal Investigator, Prof Paul Rolan, Professor Paul Rolan, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1119-9613; IBU-002 (Other: The University of Adelaide)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Medication Overuse Headache
Keywords: Medication overuse headache; ibudilast; glia
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibudilast (Experimental): To receive ibudilast 40mg twice daily for 8 weeks.
  Interventions: Drug: Ibudilast
- Placebo (Placebo Comparator): To receive placebo twice daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibudilast — Ibudilast 4 x 10 mg capsules, orally, twice daily for 8 weeks.
  Arms: Ibudilast
Drug: Placebo — Placebo 4 capsules, orally, twice daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if ibudilast is effective in reverting patients with medication overuse headache suffering chronic daily headache back to their original episodic headache pattern.

DETAILED DESCRIPTION:
It has been established that excessive intake of medications used to treat primary headaches, particularly those containing opioids, can induce a form of secondary headache, known as medication overuse headache (MOH). Despite the significant clinical impact of this condition the mechanisms behind MOH remain poorly understood, guidelines for treatment are lacking, and relapse is common.

Recently, it has been recognised that repeated opioid exposure can facilitate pain by activating glia, the immunocompetent cells of the central nervous system, resulting in opioid-induced hyperalgesia (OIH).

The investigators hypothesise that MOH represents a form of OIH in this susceptible patient group - repeated activation of nociceptive pathways by frequent headaches interacts with the opioid induced pro-inflammatory actions of activated glia to produce chronic daily headache (CDH).

This double-blind, randomised, placebo controlled pilot study will investigate the use of ibudilast, a know attenuator of glial activation, in the treatment of medication overuse headache.

ELIGIBILITY:
Inclusion criteria:

* Regular use, for at least 3 months, of opioid-containing analgesics on ≥ 10 days/month
* Headache present on at least 15 days/month, for at least 2 months
* Headache developed or markedly worsened during medication overuse
* Primary indication for analgesics is headache disorder

Exclusion criteria:

* Unable to provide written informed consent
* Age < 18 years at time of screening
* Unable to read and write in English
* Receiving tramadol regularly
* Taking triptans > 4 days/month
* Taking opioids for reasons other than headache (e.g. other pain conditions, cough, bowel motility)
* Severe psychiatric disorders
* Other chronic pain conditions likely to interfere with qualitative sensory testing (e.g. trigeminal neuralgia, arthritis)
* Diabetic neuropathy
* Recent or current active infection, determined to be clinically significant by the Principal investigator
* Known active inflammatory diseases such as rheumatoid arthritis
* History of cerebrovascular disorder
* Recent history of significant trauma, as determined by the Principal Investigator including major surgery within the previous 2 months
* Recent history of drug or alcohol abuse
* Spinal cord injury
* Any clinically significant findings on screening blood sample results
* Current malignancy
* Known hypersensitivity to ibudilast or excipients in Pinatos® formulation
* Renal or hepatic impairment, defined as baseline GFR (as calculated by the Cockcroft-Gault equation) of < 60 mL/min or LFTs > 3 times the upper limit of normal
* For females of childbearing potential:

  * Pregnancy
  * Lack of adequate contraception (abstinence, double barrier method, intrauterine device, surgical sterilization (self or partner), hormonal contraceptive methods (oral, injected, or implanted)
  * Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Headache Index | 2, 4, 8, 24 weeks
  Headache Index as calculated by the summation of headache duration (hours) X headache intensity (11-point numerical rating scale), over the final two weeks of treatment.

SECONDARY OUTCOMES:
Medication frequency | 2, 4, 8, 24 weeks
  Defined as number of days acute headache medication taken over the previous month.
Headache frequency | 2, 4, 8, 24 weeks
  Defined as number of days with headache over the previous month
Duration of headache | 2, 4, 8, 24 weeks
  Average duration of headache in hours over previous 2 weeks
Intensity of headache | 2, 4, 8, 24 weeks
  Average intensity of headache assessed by numerical rating scale over previous 2 weeks
Frequency of probable migraine attacks | 2, 4, 8, 24 weeks
  Defined as number of probable migraine attacks (using International Classification of Headache Disorders, second edition, criteria for diagnosis of migraine/migraine with aura) over previous month
Headache related impact on quality of life | 2, 4, 8, 24 weeks
  As assessed via the six-item the Headache Impact Test
Allodynia symptom checklist score | 2, 4, 8, 24 weeks
  Assesses presence of cutaneous allodynia during activities of daily living
Von Frey filament test | 2, 4, 8, 24 weeks
  To assess sensitivity to static mechanical cutaneous allodynia
Brush allodynia test | 2, 4, 8, 24 weeks
  To assess sensitivity to dynamic mechanical cutaneous allodynia
Response rate | 2, 4, 8, 24 weeks
  Response defined as ≥ 30% reduction in headache days/month or headache index from baseline. Expressed as percentage of patients who saw a ≥ 30% reduction in headache index after ibudilast treatment (at week 8) and NNT, number of patients treated to see 1 patient "respond".
Relapse rate | 2, 4, 8, 24 weeks
  Expressed as the percentage of patients who were initially classed as responders (at weeks 8) who no longer meet the criteria for responders at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rolan, MD FRACP, Principal Investigator — The University of Adelaide
Locations (1):
- Pain and Anaesthesia Research Clinic, Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Bigal ME, Lipton RB. Excessive acute migraine medication use and migraine progression. Neurology. 2008 Nov 25;71(22):1821-8. doi: 10.1212/01.wnl.0000335946.53860.1d. PMID 19029522
- [Background] Obermann M, Katsarava Z. Management of medication-overuse headache. Expert Rev Neurother. 2007 Sep;7(9):1145-55. doi: 10.1586/14737175.7.9.1145. PMID 17868013
- [Background] Hutchinson MR, Bland ST, Johnson KW, Rice KC, Maier SF, Watkins LR. Opioid-induced glial activation: mechanisms of activation and implications for opioid analgesia, dependence, and reward. ScientificWorldJournal. 2007 Nov 2;7:98-111. doi: 10.1100/tsw.2007.230. PMID 17982582